CLINICAL TRIAL: NCT00481234
Title: Heart Rate Variability for Prediction of Incidence of Cardiac Ischemia and Cardiovascular Events After General Anesthesia in High Risk Patients
Brief Title: Heart Rate Variability for Prediction of Perioperative Events
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Other Study IDs: UKSH2002_D414/02
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Anesthesia; Coronary Heart Disease
Keywords: Anesthesia, General; Abnormalities, Cardiovascular; Heart Rate; Forecasting
MeSH Terms: conditions — Coronary Disease; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Heart Rate Variability analysis

SUMMARY:
Patients with underlying cardiovascular disease are at high risk of perioperative cardiovascular events and death. Hemodynamic variables are controlled by the autonomic nervous system reflected by Heart Rate Variability. To investigate whether differences of HRV parameters predict perioperative cardiovascular events.

DETAILED DESCRIPTION:
Hypotension and bradycardia following induction of anesthesia may result in insufficient organ perfusion. Patients with underlying cardiovascular disease are at high risk of perioperative cardiovascular events and death. Hemodynamic variables are controlled by the autonomic nervous system reflected by Heart Rate Variability (HRV). Several authors demonstrated depressed long-term HRV in patients with underlying cardiovascular disease. Depressed 24 hours HRV proved to be highly predictive for cardiovascular morbidity and mortality Recently, short-term analysis was demonstrated to be a reliable tool to predict hypotension after spinal anesthesia. No data are available, however, with respect to preoperative HRV values and incidence of postoperative cardiovascular events. To investigate the prognostic value of HRV in patients with underlying cardiovascular disease. Hypothesise i) differences in pre-operative HRV are present in patients with underlying cardiovascular disease, ii) depressed preoperative HRV indicates high risk of post-operative cardiac ischemia, iii) depressed preoperative HRV is associated with longer postoperative hospital stay and adverse cardiac events after hospital discharge.

First, patients are assigned to one of two groups depending on the presence or absence of postoperative cardiac ischemia; second, a predictive model will be built to confirm our findings prospectively in another group of patients.

Patients: 100 patients (ASA physical status class II - IV) scheduled for general anesthesia. Inclusion criteria:evidence of high perioperative cardiovascular risk based on the Revised Cardiac Risk Index (RCRI >3).Exclusion criteria: lack of sinus rhythm, emergency cases, postoperative admission to an intensive care unit and age under 18 years. Time and frequency domain parameters of HRV will be recorded at the day of surgery before induction of anesthesia. Cardiovascular events and outcome will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiovascular risk factors defined as Revised Cardiac Risk Index score <= 3 scheduled for general anesthesia

Exclusion Criteria:

* Lack of sinus rhythm, emergency cases, age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2002 (Actual)
Dates: Start 2002-06; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, M.D., Prof., Principal Investigator — Chair of the Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany